CLINICAL TRIAL: NCT02824562
Title: Development of a Behavioral Intervention for Chronic Pain in Individuals With HIV
Brief Title: Pilot Testing of a Behavioral Intervention for Chronic Pain in Individuals With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jessica Merlin, MD, MBA, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: X160328007
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Other): The intervention group will receive treatment as usual plus a chronic pain self-management program which includes six one-on-one sessions facilitated by a trained interventionist and six group sessions facilitated by a trained interventionist and a peer. A peer is an HIV-infected patient living with chronic pain, who has completed all ten of the one-on-one sessions offered, received training to co-facilitate the six group sessions with the interventionist, and is successfully self-managing his/her chronic pain. The participants will complete an outcome assessment within 30 days of the last group session.
  Interventions: Behavioral: Intervention
- Control (Other): The control group will receive "treatment as usual". The "treatment as usual" or control group refers to the standard of care that patients receive for their chronic pain. This standard of care allows patients to discuss chronic pain with their providers at their discretion. Although highly variable, providers can recommend and prescribe pharmacologic (e.g., opioid and other pain medication), non-pharmacologic (e.g., physical therapy, referral to psychology) approaches for pain. This study will not interfere in any way with usual care. No additional treatment will be provided to participants allocated to the control group. The participants will complete an outcome assessment within 30 days of the last group session.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive treatment as usual plus a chronic pain self-management program which includes six one-on-one sessions facilitated by a trained interventionist and six group sessions facilitated by a trained interventionist and a peer. A peer is an HIV-infected patient living with chronic pain, who has completed all ten of the one-on-one sessions offered, received training to co-facilitate the six group sessions with the interventionist, and is successfully self-managing his/her chronic pain.
  Arms: Intervention
Behavioral: Control — The control group will receive "treatment as usual". The "treatment as usual" or control group refers to the standard of care that patients receive for their chronic pain. This standard of care allows patients to discuss chronic pain with their providers at their discretion. Although highly variable, providers can recommend and prescribe pharmacologic (e.g., opioid and other pain medication), non-pharmacologic (e.g., physical therapy, referral to psychology) approaches for pain. This study will not interfere in any way with usual care. No additional treatment will be provided to participants allocated to the control group.
  Arms: Control

SUMMARY:
Due to its specific pathophysiology and impact on health outcomes, the Institute of Medicine has described chronic pain as a complex chronic disease and a "national public health crisis." The unique neurobiological basis and psychosocial context of chronic pain in HIV-infected patients underscores the importance of developing and testing a behavioral intervention specifically tailored to this population. This study will pilot test a newly-developed behavioral intervention for chronic pain tailored to individuals with HIV.

DETAILED DESCRIPTION:
Chronic pain is a chronic condition with a unique neurobiologic basis, which has a substantial impact on physical and emotional function. Chronic pain in HIV-infected patients is common, and associated with serious health consequences, including up to 10 times greater odds of impaired physical function. Many pharmacologic therapies, including opioids, often do not lead to improved pain and function, and carry significant risk. Evidence-based behavioral interventions are among the most effective and safe non-pharmacologic chronic pain treatments investigated in the general medical population. Therefore, behavioral interventions to improve pain, physical, and emotional function in HIV-infected patients are needed. There is much to be learned from existing interventions. However, the success of a behavioral intervention is heavily influenced by how well it is tailored to the target population's biological, psychological, and social environment. Therefore, in this study investigators will conduct a two-arm pilot randomized controlled trial of a recently-developed behavioral intervention compared to routine HIV and pain care, to determine feasibility, acceptability, and preliminary impact.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Center for AIDS Research Network of Integrated Clinical Systems (CNICS) cohort
2. Age ≥ 18 years
3. Chronic pain (Brief Chronic Pain Screening Questionnaire (BCPQ) = at least moderate pain for at least 3 months)
4. Moderately severe and impairing chronic pain (PEG pain questionnaire = average of all three times is 4 or greater)

Exclusion Criteria:

1. Do not speak or understand English
2. Are planning a new pain treatment like surgery
3. Cannot attend the group sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merlin JS, Westfall AO, Johnson MO, Kerns RD, Bair MJ, Kertesz S, Turan JM, Clay OJ, Starrels JL, Kilgore M. Cost-effectiveness of a chronic pain intervention for people living with HIV (PLWH). J Med Econ. 2018 Feb;21(2):122-126. doi: 10.1080/13696998.2017.1377719. Epub 2017 Sep 18. PMID 28880698

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The intervention group will receive treatment as usual plus a chronic pain self-management program which includes six one-on-one sessions facilitated by a trained interventionist and six group sessions facilitated by a trained interventionist and a peer. A peer is an HIV-infected patient living with chronic pain, who has completed all ten of the one-on-one sessions offered, received training to co-facilitate the six group sessions with the interventionist, and is successfully self-managing his/her chronic pain.
  Behavioral intervention for chronic pain in HIV
Period: Overall Study
Arm/Group | Intervention | Control
Started | 22 | 22
Completed | 19 | 17
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [48 to 55] | 51 [46 to 57] | 51 [46 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 19 | 38
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Number of participants with undetectable viral load (blood test, measured in copies/mL) [Count of Participants; unit: Participants] | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Median Number of Study Intervention Sessions Attended by Participants
Description: Participants are expected to attend 6 one-on-one sessions and 6 group sessions. Maximum sessions if all attended per participant would be 12 sessions.
Time Frame: From baseline throughout the entire 16 week intervention period
Population: All 22 participants were assessed.
Measure: Median (Inter-Quartile Range); unit: Study Sessions
Arm/Group | Intervention
Number analyzed (Participants) | 22
Study Sessions | 9 [8 to 11]

2. Secondary Outcome: Outcome Assessment Feasibility: Number (Percentage) of Participants Who Complete Outcome Assessments Within One Month
Description: Outcome assessments are administered to participants by study staff.
Time Frame: From the conclusion of the intervention through 30 days (Intervention Group). From the last group session through 30 days (Control Group).
Population: All 22 participants in each arm were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22 | 22
Participants
  Completed outcome assessment | 19 | 17
  Did not complete outcome assessment | 3 | 5

ADVERSE EVENTS:
Time Frame: During the intervention phase of the study, up to 16 weeks from the first group session
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT02824562/Prot_SAP_000.pdf